CLINICAL TRIAL: NCT06773182
Title: Understanding Patient's Barriers and Perceived Benefits Through Adherence to Nutritional Interventions in IBD: a Preliminary Study.
Brief Title: Assessing Interventions of Diet in IBD
Acronym: AID-IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, David Armstrong, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB #18028
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: IBD (Inflammatory Bowel Disease); Ulcerative Colitis (UC); Crohn Disease (CD)
Keywords: IBD; Low FODMAP Diet; Mediterranean diet; Intermittent fasting; Ulcerative colitis; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This is a mixed-design, randomized, parallel-group trial with three independent arms. Participants will be randomly assigned to one of three dietary intervention groups: intermittent fasting, the Mediterranean diet, or the Low FODMAP diet. Each arm will operate independently, and participants will adhere exclusively to their assigned dietary intervention throughout the study duration. The design ensures that the effects of each diet are evaluated in isolation, allowing for a direct comparison of adherence rates, perceived benefits, and impacts on IBD symptom management across the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Fasting (Experimental): Participants will be assigned to follow an intermittent fasting protocol.
- Mediterranean Diet (Experimental): Participants will be assigned to follow a Mediterranean diet.
- Low FODMAP Diet (Experimental): Participants will be assigned to follow a Low FODMAP Diet.
  Interventions: Other: Low FODMAP Diet Intervention

INTERVENTIONS:
Other: Intermittent Fasting Intervention — A 14:10 intermittent fasting regimen, where participants fast for 14 hours and consume all meals within a 10-hour eating window daily.
Other: Mediterranean Diet Intervention — A diet emphasizing whole grains, fruits, vegetables, olive oil, lean proteins, and minimizing processed foods.
Other: Low FODMAP Diet Intervention — A diet limiting fermentable oligosaccharides, disaccharides, monosaccharides, and polyols to manage gastrointestinal symptoms.
  Arms: Low FODMAP Diet

SUMMARY:
In this study, we are trying to learn how certain diets affect people with inflammatory bowel disease (IBD). We want to understand what makes it hard or easy for them to stick to different eating plans, like intermittent fasting, the Mediterranean diet, and the Low FODMAP diet. By finding out how these diets help with symptoms and which ones are easier to follow, we hope to improve the quality of life for people with IBD.

DETAILED DESCRIPTION:
This study aims to explore the impact of specific dietary interventions on individuals living with inflammatory bowel disease (IBD). By examining dietary patterns such as intermittent fasting, the Mediterranean diet, and the Low FODMAP diet, we seek to identify barriers to adherence and facilitators that make these eating plans sustainable. Additionally, we aim to evaluate the perceived benefits of these diets in managing IBD symptoms and their influence on overall quality of life. The findings will provide valuable insights to develop patient-centered nutritional strategies that enhance adherence and therapeutic outcomes in IBD care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years) diagnosed with ulcerative colitis or Crohn's disease.
* Having willingness to use their personal smartphone to access the app
* Able to understand the indication by the registered dietitian.
* Able to provide informed consent.
* Willingness to attempt intervention diet and commit to study procedures.

Exclusion Criteria:

* Pregnant women.
* Currently being treated for eating disorders, schizophrenia, psychosis, or other acute mental disorders.
* Currently being treated for chemotherapy.
* Diabetes
* Advance chronic kidney disease
* Short bowl syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To identify IBD's top three patients' barriers to access and follow the nutritional intervention. | From enrollment to the end of the study and at 5 weeks
  The outcome will be assessed through semi-structured one-on-one interviews conducted at the end of the study. Interviews will last approximately 40 minutes to 1 hour and will follow a structured interview guide with open-ended questions, designed to explore participants' experiences, perceptions, and challenges in accessing and adhering to the nutritional intervention. Interviews will be audio-recorded and transcribed verbatim.
  Data will be analyzed using thematic analysis informed by interpretive description methodology, to identify key personal and systemic barriers. NVivo software (QSR International) will be used to facilitate qualitative coding and analysis.

SECONDARY OUTCOMES:
To identify specific sociodemographic criteria that may act as a deterrent or facilitator in the ability to generate honest qualitative data through questionnaires and an individual interview. | From enrollment to the end of the study and at 5 weeks
To identify adherence to each food intervention through the use of an app (RxFood) and different questionnaires. | From enrollment to the end of the study and at 5 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - 2F Digestive Diseases Clinic - Hamilton Health Science, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Approach investigators to ask for anonymized dataset
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after data completion - estimated 1 year
Access Criteria: The research team who will evaluate the interventions of diet in IBD